CLINICAL TRIAL: NCT00725686
Title: A Phase I Open-Label, Dose Escalation Trial Of REDD14NP Delivered By A Single Intravitreal Injection To Patients With Choroidal Neovascularization (CNV) Secondary To Exudative Age-Related Macular Degeneration ("Wet AMD").
Brief Title: Study of PF-04523655 (REDD14NP) In Subjects With Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (Wet AMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quark Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B0451008; QRK.003 (Other: Quark Pharmaceuticals Inc.); NCT00455481 (obsolete NCT alias)
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Age-Related Macular Degeneration
Keywords: Choroidal Neovascularization (CNV) "WET" AMD
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — PF-04523655

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PF-04523655 — This is a dose-escalation study (50, 100, 200, 400, 670, 1000, 1500, 2250, 3000 microgram) given at baseline and then the subject is followed up for 24 months
  Other Names: REDD14NP

SUMMARY:
The aim of the study is to evaluate whether PF-04523655 is safe in the treatment of neovascular/wet AMD

DETAILED DESCRIPTION:
Dose escalation safety study

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 50 years old and in general good health. Patients with medically controlled chronic disease such as HTN, AODM, and hyperlipidemia may be included.
* Patient is capable of giving consent.
* Patient is willing and able to comply with the visit schedule and study procedures including follow-up visits.
* Patient has documented CNV secondary to AMD with evidence of active disease characterized by blood vessel leakage or evidence of hemorrhage.
* Patient has clear ocular media and adequate pupil dilation to allow good quality imaging by fundus photography.
* Patient's intraocular pressure is ≤ 25 mmHg

Exclusion Criteria:

* Patient is of childbearing potential. Every female patient is considered of child-bearing potential unless she has had sterilization surgery or is post-menopausal and has not had a menstrual period for at least 12 months.
* Patient has CNV due to causes other than AMD, including ocular or periocular infections.
* Patient has lesions not easily imaged and quantified.
* Patient has underlying systemic disease such as cardiac, neurological, infectious disease, uncontrolled diabetes mellitis, or disease of the eye other than AMD. Patient may have medically controlled glaucoma.
* Patient is participating in any concurrent interventional study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of PF-04523655 when administered as a single intravitreal injection | Over a 24-Month Period

SECONDARY OUTCOMES:
To describe anatomical changes in the retina and choroid following the administration of PF-04523655 | Day 14
To determine the changes in visual acuity ETDRS chart after a single intravitreal injection of PF-04523655 | Day 14
To evaluate the safety, efficacy and frequency of dosing following administration of PF-04523655 of approved VEGF-inhibitors in those study patients requiring rescue therapy | Monthly
To evaluate early response after a single intravitreal administration of PF-04523655 in patients who, in the opinion of the investigator, have the potential to show improvement in visual acuity from other treatment options (Stratum 2 patients) | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (8):
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, ‘Aiea, Hawaii
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio
- Israel (3):
  - Pfizer Investigational Site, Tel Aviv, Israel
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Rehovot

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0451008&StudyName=A%20Phase%201%20Dose%20Escalation%20Study%20of%20PF-04523655%20%28REDD14NP%29%20In%20Subjects%20with%20Choroidal%20Neovascularization%20%28CNV%29%20Secondary%20to%20Age-Relat